CLINICAL TRIAL: NCT04928781
Title: Smoking Cessation Intervention for Hospitalized Heart & Vascular Center (HVC) Patients at a Dartmouth-Hitchcock Medical Center Serving a Rural Population
Brief Title: Smoking Cessation Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI and funding source collectively decided to close study due to lack of smoking cessation counselor required for study
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Merle L. Myerson, Staff Physician, Cardiovascular Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02000943
Record Dates: First submitted 2021-06-02; First posted 2021-06-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Smoking Cessation
Keywords: Percutaneous Coronary Intervention
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: 2 arm study, with a control arm and intervention arm. The control arm will consist of a retrospective chart review will be conducted to create a randomly selected cohort of patients that meet inclusion and exclusion criteria and did not receive smoking cessation counseling to serve as the control arm. The intervention arm will prospectively enroll to be provided with smoking cessation counseling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking Cessation Counseling - Intervention Arm (Experimental): Intervention arm. All patients enrolled in the study will be provided with smoking cessation counseling.
  Interventions: Behavioral: Smoking Cessation Counseling
- Retrospective Chart Review - Control Arm (No Intervention): Control arm. A retrospective chart review will be conducted to create a randomly selected cohort of patients that meet inclusion and exclusion criteria and did not receive smoking cessation counseling to serve as the control arm.

INTERVENTIONS:
Behavioral: Smoking Cessation Counseling — Smoking cessation counseling will be provided following standards set by the institution patients are receiving care at (Dartmouth-Hitchcock Medical Center).
  Arms: Smoking Cessation Counseling - Intervention Arm

SUMMARY:
This is a pilot study to determine the feasibility and success of offering smoking cessation counseling for ambulatory patients who present for scheduled cardiac catheterization.

DETAILED DESCRIPTION:
This is a prospective randomized pilot study of feasibility and success of smoking cessation counselling for ambulatory patients who present for scheduled cardiac catheterization. Patients who meet inclusion and exclusion criteria will be eligible for enrollment and receive smoking cessation counseling. Patients will be followed for 6 months post intervention. A Usual care arm will be created using retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* Presents to Dartmouth-Hitchcock Medical Center in Lebanon, NH as an ambulatory patient with a scheduled cardiac Catheterization
* smoke one or more cigarettes per day for the past 12 months OR use of electronic-cigarettes containing tobacco at least once during the past 30 days.
* proficient in English

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-28 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants that self-report sustained smoking cessation | 1 month post index procedure
  Percentage of participants that self report sustained smoking cessation at 1 month.
Percentage of participants that self-report sustained smoking cessation | 3 months post index procedure
  Percentage of participants that self report sustained smoking cessation at 3 months.
Percentage of participants that self-report sustained smoking cessation | 6 months post index procedure
  Percentage of participants that self report sustained smoking cessation at 6 months.

SECONDARY OUTCOMES:
Percentage of participants that have had at least one subsequent cardiovascular hospital admission. | 1 month post index procedure
  Percentage of participants that have had at least one subsequent cardiovascular hospital admission at 1 month post index procedure.
Percentage of participants that have had at least one subsequent cardiovascular hospital admission. | 3 months post index procedure
  Percentage of participants that have had at least one subsequent cardiovascular hospital admission at 3 months post index procedure.
Percentage of participants that have had at least one subsequent cardiovascular hospital admission. | 6 months post index procedure
  Percentage of participants that have had at least one subsequent cardiovascular hospital admission at 6 months post index procedure.
Percentage of participants that have had at least one emergency department presentation | 1 month post index procedure
  Percentage of participants that have had at least one emergency department presentation following discharge for their index procedure 1 month post index procedure
Percentage of participants that have had at least one emergency department presentation | 3 months post index procedure
  Percentage of participants that have had at least one emergency department presentation following discharge for their index procedure 3 months post index procedure
Percentage of participants that have had at least one emergency department presentation | 6 months post index procedure
  Percentage of participants that have had at least one emergency department presentation following discharge for their index procedure 6 months post index procedure
Frequency of Cardiac Events following discharge from index procedure | 1 month post index procedure
  Frequency of cardiac events following discharge from hospitals, 1 month after index procedure.
Frequency of Cardiac Events following discharge from index procedure | 3 months post index procedure
  Frequency of cardiac events following discharge from hospitals, 3 months after index procedure.
Frequency of Cardiac Events following discharge from index procedure | 6 months post index procedure
  Frequency of cardiac events following discharge from hospitals, 6 months after index procedure.
Percentage of participants that need subsequent coronary intervention following index procedure | 1 month post index procedure
  Percentage of participants that need subsequent coronary intervention following index procedure at 1 month post index procedure
Percentage of participants that need subsequent coronary intervention following index procedure | 3 moths post index procedure
  Percentage of participants that need subsequent coronary intervention following index procedure at 3 months post index procedure
Percentage of participants that need subsequent coronary intervention following index procedure | 6 months post index procedure
  Percentage of participants that need subsequent coronary intervention following index procedure at 6 months post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Merle L Myerson, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Health, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
No Plant to share individual participant data (IPD) exists at this time.